CLINICAL TRIAL: NCT04623177
Title: Effectiveness of Thromboprophylaxis With Low Molecular Weight Heparin in Critically Ill Patients With COVID-19. A Prospective, Cohort, Multicenter Study.
Brief Title: Thromboprophylaxis for Patients in ICU With COVID-19
Status: Completed | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Hospital Universitario Doctor Peset (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario La Paz (Other); Hospital Universitario La Fe (Other); Hospital de Sant Joan Despí Moisès Broggi (Other); University of Navarrra Hospital (Clinica Universitaria) (Other); Hospital de Cruces (Other)
Responsible Party: Sponsor
Other Study IDs: RegCoVid-19
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-10

CONDITIONS: Covid19; Anticoagulant Therapy; Thrombosis
Keywords: Covid19; Low Molecular weight heparin; Thromboprophylaxis; Anticoagulant treatment; Thrombosis
MeSH Terms: conditions — COVID-19; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anticoagulation: Patients receiving an anticoagulant dose (equal or higher than 150 IU/kg/24 h) of LMWH within the first 48 hours after the ICU admission
- Thromboprophylaxis: Patients receiving a prophylactic dose (lower than 150 IU/kg/24 h) of LMWH within the first 48 hours after the ICU admission
- No heparin: Patients receiving no anticoagulant drug within the first 48 hours after the ICU admission

SUMMARY:
The respiratory distress that goes with COVID-19 infection has been related to a procoagulant state, with thrombosis at both venous and arterial levels, that determines hypoxia and tissue dysfunction at several organs. The main sign of this thrombotic activity seems to be the D-Dimers, that have been proposed to identify patients with poor prognosis at an early stage.

Knowledge on how to prevent or even treat this procoagulant state is scarce. COVID-19 patients may be out of general thromboprophylaxis recommendations, and recent studies suggest a better prognosis in severe COVID-19 patients receiving anticoagulant therapy with low molecular weight heparin (LMWH). However, the LMWH efficacy and safety, mainly in patients admitted to an Intensive Care Unit, remains to be validated.

DETAILED DESCRIPTION:
Many reports have postulated a procoagulant state along with the respiratory distress caused by coronavirus SARS-CoV2. A complex physiopathology has been proposed trying to explain this profile, mainly based on the thromboinflammatory concept, with thrombosis at both venous and arterial levels. Microvascular thrombi impair the blood flow all over the body, with a vascular shunt due to capillary obstruction, that determines hypoxia and tissue dysfunction at several organs, being the lung the more affected one.

Although D-Dimers (DD) are not specific indicators of clot formation, its elevation, in combination with other parameters (hyperfibrinogenemia, mild thrombocytopenia) may suggest a systemic coagulation activation with an increase of thrombin generation and fibrinolysis. In fact, in a retrospective Chinese analysis, a DD higher than 1000 ng/ml was proposed to identify patients with poor prognosis at an early stage.

Nevertheless, knowledge on how to prevent or even treat this procoagulant state is scarce. Thromboprophylaxis with low molecular-weight heparin (LMWH) is recommended in most medical patients admitted to the hospital and in nearly all patients in an Intensive Care Unit (ICU). But COVID-19 patients may be out of these recommendations, and some treatment schemes has been proposed, although how to decide the suitable LMWH for each clinical situation is controversial. Recent retrospective studies suggest a better prognosis in severe COVID-19 patients receiving anticoagulant therapy with LMWH. However, the LMWH efficacy and safety, mainly in COVID-19 patients admitted to the ICU, remains to be validated.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV2 infection from a respiratory tract sample using a polymerase chain reaction assay.
* Admitted to ICU

Exclusion Criteria:

* Non-confirmed SARS-CoV2 infection
* No data at first day ICU admission
* Patient with do-not resuscitate orders
* Patient who did not meet the outcomes of death or ICU discharge by the time of study completion date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive COVID-19 patients admitted to participating ICUs from March 12th to September 1st were included if they fulfill the inclusion criteria and present no exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 822 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
ICU mortality | From admission to ICU discharge, an average of 1 month
  Rate of mortality

SECONDARY OUTCOMES:
ICU incidence of thrombotic events | From admission to ICU discharge, an average of 1 month
  A composite endpoint to evaluate efficacy made up of: myocardial infarction, stroke, incidental pulmonary thromboembolism, pulmonary thromboembolism with worsening of hypoxemia, Pulmonary thromboembolism with hemodynamic repercussion, other venous thromboses without pulmonary thromboembolism
ICU incidence of bleeding events | From admission to ICU discharge, an average of 1 month
  Composite endpoint to evaluate safety made up of: bleeding needing transfusion, bleeding wit hemodynamic repercussion, other bleeding (minor bleeding)
Length of ICU stay | From admission to ICU discharge, an average of 1 month
  Days admitted in ICU
Length of invasive mechanical ventilation | From admission to ICU discharge, an average of 1 month
  Days treated with invasive mechanical ventilation (controlled or assisted)
Effect of LMWH in other parameters | From admission to ICU discharge, an average of 1 month
  Description of the relationship if any between the use of LMWH and thrombotic or inflammatory parameters (D-Dimer levels, ferritin) or lung dead space

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Ferrandis, MD, Study Chair — Hospital Universitario La Fe
Locations (31):
- Spain (31):
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario de Araba, Álava, Basque Country
  - Complejo Asistencial Universitario de León, León, Castille and León
  - Hospital Universitario Rio Ortega, Valladolid, Castille and León
  - Hospital General de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Hospital Clinic Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital de Terrasa, Barcelona, Catalonia
  - Complejo Hospitalario de Cáceres, Cáceres, Extramedura
  - Hospital Unversitario A Coruña, A Coruña, Galicia
  - Complexo Hospitalario Universitario de Ferrol, A Coruña, Galicia
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra, Galicia
  - Hospital Povisa, Pontevedra, Galicia
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas, Gran Canaria
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Universitario San Juan de Alicante, Alicante, Valencia
  - Hospital del Mar, Barcelona
  - Hospital Sanitas Cima, Barcelona
  - Hospital Sant Joan Despí, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Infanta Sofia, Madrid
  - Hospital Rafael Méndez, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitari La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Jackson SP, Darbousset R, Schoenwaelder SM. Thromboinflammation: challenges of therapeutically targeting coagulation and other host defense mechanisms. Blood. 2019 Feb 28;133(9):906-918. doi: 10.1182/blood-2018-11-882993. Epub 2019 Jan 14. PMID 30642917
- [Background] Ferrandis R, Llau JV, Quintana M, Sierra P, Hidalgo F, Cassinello C, Gomez-Luque A. COVID-19: opening a new paradigm in thromboprophylaxis for critically ill patients? Crit Care. 2020 Jun 11;24(1):332. doi: 10.1186/s13054-020-03052-9. No abstract available. PMID 32527286
- [Background] Llau JV, Ferrandis R, Sierra P, Hidalgo F, Cassinello C, Gomez-Luque A, Quintana M, Amezaga R, Gero M, Serrano A, Marcos P. SEDAR-SEMICYUC consensus recommendations on the management of haemostasis disorders in severely ill patients with COVID-19 infection. Rev Esp Anestesiol Reanim (Engl Ed). 2020 Aug-Sep;67(7):391-399. doi: 10.1016/j.redar.2020.05.007. Epub 2020 May 23. PMID 32591185
- [Background] Paranjpe I, Fuster V, Lala A, Russak AJ, Glicksberg BS, Levin MA, Charney AW, Narula J, Fayad ZA, Bagiella E, Zhao S, Nadkarni GN. Association of Treatment Dose Anticoagulation With In-Hospital Survival Among Hospitalized Patients With COVID-19. J Am Coll Cardiol. 2020 Jul 7;76(1):122-124. doi: 10.1016/j.jacc.2020.05.001. Epub 2020 May 6. No abstract available. PMID 32387623
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Tang N, Bai H, Xiong D, Sun Z. Specific coagulation markers may provide more therapeutic targets in COVID-19 patients receiving prophylactic anticoagulant. J Thromb Haemost. 2020 Sep;18(9):2428-2430. doi: 10.1111/jth.14988. No abstract available. PMID 32619329
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112